CLINICAL TRIAL: NCT01645332
Title: Role of DLBS3233 in the Treatment of Subjects With New Onset of Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of DLBS3233 in Subjects With New Onset of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS3233-0912
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Type-2-diabetes Mellitus; New Onset
Keywords: DLBS3233; new onset; type-2-diabetes mellitus; oral anti-hyperglycemic agent
MeSH Terms: interventions — DLBS3233

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment I (control) (Placebo Comparator): Placebo of DLBS3233 once daily for 12 weeks + lifestyle modification
  Interventions: Drug: Placebo of DLBS3233; Other: Lifestyle modification
- Treatment II (Experimental): 100 mg DLBS3233 once daily for 12 weeks + lifestyle modification
  Interventions: Drug: DLBS3233; Other: Lifestyle modification

INTERVENTIONS:
Drug: Placebo of DLBS3233 — Placebo of DLBS3233 once daily for 12 weeks
  Other Names: Placebo of Inlacin
  Arms: Treatment I (control)
Drug: DLBS3233 — 100 mg DLBS3233 once daily for 12 weeks
  Other Names: Inlacin
  Arms: Treatment II
Other: Lifestyle modification — Each study subject will be provided with and instructed to follow a lifestyle modification (particularly regarding dietary advice and exercise) during the subject's participation in the study.

SUMMARY:
This is a 2-arm, double-blind, parallel, randomized, placebo-controlled clinical study, with 12 weeks of therapy to evaluate the efficacy and safety of DLBS3233 in improving metabolic control in newly diagnosed type-2-diabetic patients, as measured by A1c level, fasting and 2-hours post-prandial plasma glucose, fasting insulin level, HOMA-IR, HOMA-B, adiponectin level, lipid profile, and body weight.

DETAILED DESCRIPTION:
There will be two groups of treatment in this study who will receive DLBS3233 or placebo of DLBS3233 (with lifestyle modification) for 12 weeks of therapy.

Clinical and physical examination to evaluate the efficacy and safety as well as measurement of fasting and 2-hour post-prandial plasma glucose level will be performed at baseline and every 6-weeks-interval. Other clinical and laboratory examinations will be performed at baseline and at the end of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age of 18-60 years
* BMI ≥ 18.5 kg/m2
* Newly diagnosed (new onset of) type 2 DM subjects, defined as FPG level of ≥ 126 mg/dL or 2h-PG level of ≥ 200 mg/dL or A1c of ≥ 6.5%)
* FPG ≤ 183 mg/dL
* Hemoglobin level of ≥ 10.0 g/dL
* Serum ALT ≤ 2.5 times upper limit of normal
* Serum creatinine < 1.5 times upper limit of normal

Exclusion Criteria:

* Female of childbearing potential
* Subjects with symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or other symptomatic ischemic arterial diseases necessitating medical treatment
* Uncontrolled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg)
* History of renal and/or liver disease
* History of or the presence of any clinical evidence of malignancies
* Presence of exacerbation of chronic illnesses, severe and acute infections, complicated infections
* Current treatment with systemic corticosteroids or herbal (alternative) medicines
* Participation in any other intervention trial within 30 days prior to Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Reduction of A1c level | 12 weeks
  Reduction of A1c level from baseline to Week 12 of treatment

SECONDARY OUTCOMES:
Reduction of venous FPG | 6 weeks and 12 weeks
  Reduction of venous FPG from baseline to Week 6 and Week 12 of treatment
Reduction of venous 2h-PG | 6 weeks and 12 weeks
  Reduction of venous 2h-PG from baseline to Week 6 and Week 12 of treatment
Response rate | 12 weeks
  Percentage of subjects with FPG < 110 mg/dL and/or reduction of at least 10% in FPG level from baseline to Week 12 of treatment
Change in fasting insulin level | 12 weeks
  Change in fasting insulin level from baseline to Week 12 of treatment
Change in HOMA-IR | 12 weeks
  Change in HOMA-IR from baseline to Week 12 of treatment
Change in HOMA-B | 12 weeks
  Change in HOMA-B from baseline to Week 12 of treatment
Change in adiponectin level | 12 weeks
  Change in adiponectin level from baseline to Week 12 of treatment
Change in lipid profile | 12 weeks
  Change in lipid profile (LDL-cholesterol, HDL-cholesterol, total cholesterol, and triglyceride levels) from baseline to Week 12 of treatment
Change in body weight | 6 weeks and 12 weeks
  Change in body weight from baseline to Week 6 and Week 12 of treatment
Vital signs | 6 weeks and 12 weeks
  Vital signs (blood pressure, heart rate, respiratory rate) will be measured at baseline, Week 6, and Week 12
Liver function | 12 weeks
  Liver function (serum ALT, serum AST, serum γ-glutamyl transferase levels) will be evaluated at baseline and Week 12
Renal function | 12 weeks
  Renal function (serum creatinine level) will be evaluated at baseline and Week 12
Electrocardiography (ECG) | 12 weeks
  ECG will be evaluated at baseline and Week 12
Adverse events | 12 weeks
  Adverse events as well as number of subjects experienced the events will be observed and evaluated throughout study period (12 weeks) and until all adverse events have been recovered or stabilized

CONTACTS AND LOCATIONS:
Overall Officials: Heri Nugroho, Dr,dr,SpPD,KEMD,FINASIM, Principal Investigator — Division of Endocrinology, Department of Internal Medicine, Faculty of Medicine, Diponegoro University, Dr. Kariadi Hospital, Semarang, Indonesia
Locations (1):
- Division of Endocrinology, Department of Internal Medicine, Dr. Kariadi Hospital, Semarang, Central Java, Indonesia